CLINICAL TRIAL: NCT06329765
Title: CUped: An Approach to Motor Recovery Post-Stroke, Not Compensation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sheila Schindler-Ivens, Associate Professor, Marquette University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR- 4380
Record Dates: First submitted 2023-10-06; First posted 2024-03-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single group pretest-posttest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise with CUped (Experimental): Participants will exercise with CUped (a motor-assisted, split crank pedaling device) and undergo 50 m of gait training. CUped comprises a left and right pedal; each is attached to the shaft of a motor. There is no mechanical connection between pedals. Participant's feet are secured to the pedals. They are asked to pedal forward and keep the legs 180° out-of-phase. The position of the left and right cranks is monitored. When the phase relationship is not maintained, motors provide torque to assist the lagging limb and resist the leading limb. Motors are under feedback control. Torque is proportional to the magnitude and sign of the error.
  Interventions: Behavioral: Exercise with CUped - a motor-assisted, split crank pedaling device and undergo 50 m of gait training.

INTERVENTIONS:
Behavioral: Exercise with CUped - a motor-assisted, split crank pedaling device and undergo 50 m of gait training. — Exercise with CUped - a motor-assisted, split crank pedaling device and undergo 50 m of gait training.
  Other Names: Exercise with CUped

SUMMARY:
The goal of lower limb rehabilitation after stroke is recovery of independent walking at home and in the community. Few stroke survivors achieve this goal. Suboptimal outcomes are due to the serious and intransigent nature of movement impairments caused by stroke and the scarcity of feasible and effective therapies that restore movement lost to stroke. Our team has developed a novel exercise intervention called CUped (pronounced cupid, like the Roman god) to address barriers to recovery and improve walking after stroke. CUped is so called because it compels use of the paretic limb during a movement that resembles pedaling. This project will examine safety, acceptability, and tolerance to CUped, characterize its therapeutic effects, and identify dose-response relationships. Results will provide preliminary data for an R01 to support a randomized controlled trial (RCT). CUped is designed to help stroke survivors recover lower limb movement lost to stroke, thereby improving walking. It is intended to be used as an adjunct to gait training. CUped uses a robotic technology that eliminates compensatory movements that interfere with recovery, compels use of the paretic lower limb, and targets 3 key movement impairments caused by stroke: decreased muscle output from the paretic limb, inappropriate paretic muscle timing, and abnormal interlimb coordination. Exercise is done in sitting which enables high repetition practice. Like walking, CUped requires continuous, reciprocal use of both lower limbs; effects are likely to transfer to walking. The risk-reward profile of this proposal is ideal for an R21, which is an NIH funding opportunity intended to encourage exploratory/developmental research by providing support for the early and conceptual stages of project development. CUped is a novel therapy grounded in a physiologic premise and based on prior observations from our laboratory. The investigators have pilot data suggesting that CUped fulfills its design specifications, and this study will be the first to test its therapeutic effects. In this Stage 1 rehabilitation trial, The investigators will support or quickly refute the hypothesis that CUped is safe, acceptable, and capable of eliciting a therapeutic response in stroke survivors. The investigators will also examine tolerance to CUped and dose-response effects. If our hypotheses are supported, the investigators will be poised to run an RCT to isolate the effects of CUped and compare them to standard care. Future work will investigate physiologic mechanisms underlying the effects of CUped.

DETAILED DESCRIPTION:
The goal of lower limb rehabilitation after stroke is recovery of independent walking at home and in the community. Few stroke survivors achieve this goal. Suboptimal outcomes are due to the serious and intransigent nature of movement impairments caused by stroke and the scarcity of feasible and effective therapies that restore movement lost to stroke. Our team has developed a novel exercise intervention called CUped (pronounced cupid, like the Roman god) to address barriers to recovery and improve walking after stroke. CUped is so called because it compels use of the paretic limb during a movement that resembles pedaling. This project will examine safety, acceptability, and tolerance to CUped, characterize its therapeutic effects, and identify dose-response relationships. Results will provide preliminary data for an R01 to support a randomized controlled trial (RCT). CUped is designed to help stroke survivors recover lower limb movement lost to stroke, thereby improving walking. It is intended to be used as an adjunct to gait training. CUped uses a robotic technology that eliminates compensatory movements that interfere with recovery, compels use of the paretic lower limb, and targets 3 key movement impairments caused by stroke: decreased muscle output from the paretic limb, inappropriate paretic muscle timing, and abnormal interlimb coordination. Exercise is done in sitting which enables high repetition practice. Like walking, CUped requires continuous, reciprocal use of both lower limbs; effects are likely to transfer to walking. The risk-reward profile of this proposal is ideal for an R21. CUped is a novel therapy grounded in a physiologic premise and based on prior observations from our laboratory. The investigators have preliminary data suggesting that CUped fulfills its design specifications, and this study will be the first to test its therapeutic effects. In this Stage 1 rehabilitation trial, the investigators will support or quickly refute the hypothesis that CUped is safe, acceptable, and capable of eliciting a therapeutic response in stroke survivors. The investigators will also examine tolerance to CUped and dose-response effects. If our hypotheses are supported, the investigators will be poised to run an RCT to isolate the effects of CUped and compare them to standard care. Future work will investigate physiologic mechanisms underlying the effects of CUped. CUped uses a split-crank pedaling apparatus with no mechanical connection between the right and left pedals. Participants are asked to pedal with both limbs while maintaining a 180° phase relationship. When appropriate phasing is not maintained, motors assist the lagging limb and resist the leading limb until the desired phasing is restored. CUped can also be configured for unilateral and conventional coupled pedaling. Stroke survivors will be asked to participate in 24 exercise sessions with CUped. They will be encouraged to perform up to 12 bouts of bilateral uncoupled (i.e., split-crank) pedaling with motorized intervention. Exercise will continue until all 12 bouts have been completed or the task cannot be sustained. Immediately after exercising with CUped, participants will perform 1 bout of overground gait training. Safety, acceptability, tolerance, and movement ability will be assessed to examine the following specific aims: Aim 1: Establish safety, acceptability, and tolerance to CUped. During training, the investigators will track adverse events, absences, and the number of repetitions per session of bilateral uncoupled pedaling (reps/session). If there are no adverse events related to participation, the investigators will conclude that CUped is safe. If ≥75% of participants attend ≥75% of training sessions, the investigators will conclude that the intervention is acceptable. Reps/session will be used to quantify tolerance, which is expected to increase across sessions. As one measure of exercise dose, tolerance will be used to characterize dose-response relations and to develop a training protocol for an RCT. Safety, acceptability, and patient tolerance are preconditions of an RCT, and they are imperative for clinical adoption. Clinical impact demands safe and effective interventions that are feasible and readily accepted by the target population. Aim 2: Characterize therapeutic responses to CUped and their relationship to dose. Paretic limb use and interlimb coordination will be assessed before, after, and at the midpoint of training. Measures will be made during walking and pedaling. An ideal result would be significant improvement in paretic limb use and interlimb coordination during walking. However, this outcome relies on task-specific effects in pedaling that transfer to walking. Hence, improved pedaling performance and decreased use of motorized intervention will be assessed for evidence of intermediate effects. Correlation will be used to examine relationships between therapeutic responses and exercise dose. Measures with significant correlations will be used to develop a regression model describing dose-response relations and to establish dosing protocols.

ELIGIBILITY:
Inclusion Criteria:

* Single, unilateral stroke in adulthood.
* Cortical, subcortical stroke. Individuals with cortical lesions affecting sensory and motor structures in the gray matter of the brain will be included. Individuals subcortical white matter lesions affecting the internal capsule and corona radiata will be included.
* Ischemic, hemorrhagic stroke. Individuals with ischemic and hemorrhagic strokes will be admitted. Because ischemic stroke is more common than hemorrhagic, the investigators expect a smaller proportion of volunteers from the latter group.
* Chronic stroke. Individuals with chronic stroke, deﬁned as >6 months post infarct, will be included.
* Able to walk 10 m. Stroke survivors capable of walking 10 m overground will be admitted. Canes, walkers, braces, and other devices will be allowed. This study examines the effect of CUped on gait kinematics and kinetics; therefore, the ability to walk is imperative.
* Unilateral motor impairment consistent with hemiparesis.
* Learned non-use of the paretic limb. Non-use will be veriﬁed by comparing paretic limb work (W) during unilateral and bilateral coupled pedaling. Participants with non-use will be identiﬁed as those who produce signiﬁcantly <50% of the total W of bilateral coupled pedaling with their paretic limb but are capable of unilateral pedaling with the paretic limb at a workload equivalent to 50% of the total W of bilateral coupled pedaling. (Signiﬁcance will be determined using a 1-sample t-test or corresponding non-parametric test in the case of non-normality).
* No contraindications for exercise. Contraindications to exercise include but may not be limited to recent electrocardiogram changes or recent myocardial infarction, uncontrolled arrhythmia, unstable angina, third degree heart block, acute progressive heart failure, uncontrolled hypertension, and orthopedic conditions (e.g., severe muscle contracture, arthritis, acute limb injury) that may interfere with pedaling.
* Age ≥18. All participants must be at least 18 years of age. The investigators are studying adult not childhood stroke. Recovery mechanisms are different between adult and childhood stroke survivors.
* Able to commit to 27 visits to the lab (pre-, mid-, post-test, plus 24 training sessions).

Exclusion Criteria:

* More than 1 stroke. Individuals with more than one clinically apparent stroke, as evidenced by residual impairments and/or medical imaging, will be excluded. Individuals with history of transient ischemic attack (TIA) resulting in no residual impairments or brain damage will NOT be excluded.
* Stroke in the cerebellum or basal ganglia. Individuals with stroke affecting primarily the cerebellum or basal ganglia will be excluded. The cerebellum has an important role in motor learning. Given that CUped depends on motor learning, people with cerebellar strokes may not beneﬁt. Basal ganglia strokes can cause tremor, which is not the target of CUped. However, individuals with predominantly internal capsule lesions that also affect the basal ganglia will be included.
* Dementia or other cognitive impairment that interferes with learning and/or the ability to consent.
* Communication impairments, such as receptive aphasia, that prevent safe participation. Expressive aphasia is not an exclusion criterion. Participants will be included as long as they have a method to communicate willingness to participate, discomfort, and/or the desire to start or stop a study activity.
* Orthopedic impairments that interfere with pedaling.
* Cardiovascular contraindications to exercise.
* Inability to walk 10 m overground. Participants will be excluded in they are not able to walk 10 m overground our cannot do so safely.
* Neurological disorder other than stroke. Individuals with history or signs of any neurologic disease or injury other than stroke will be excluded. Such conditions may include head trauma, cerebral palsy, epilepsy, brain tumor, diabetic neuropathy, dementia, multiple sclerosis, Parkinson's disease, or Alzheimer's disease.
* Other conditions that interfere with safe participation or data integrity. Participants will be excluded if, at any point in the recruitment or enrollment process, the investigators become aware of a condition that increases risk beyond that indicated in our IRB protocols. Exclusion will also occur if the investigators become aware of a condition that introduces an experimental variable that could confound the results of the study.
* Failure to meet any inclusion criteria listed above.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2027-04-04 (Estimated)

PRIMARY OUTCOMES:
Paretic limb use in walking | Pretest (1 day to 1 month before the intervention begins), Posttest (typically within 1 week of completing the intervention) and Midpoint of training (week 3)
  Propulsive impulse generated by the paretic limb during overground walking measured from biomechanical gait analysis.
Paretic limb use in pedaling | Each training day, up to 24 times, through study completion which takes 6-8 weeks.
  Mechanical work generated by the paretic limb during conventional pedaling measured from force-sensitive pedals.
Interlimb coordination in walking | Pretest (1 day to 1 month before the intervention begins), Posttest (typically within 1 week of completing the intervention) and Midpoint of training (week 3)
  Interlimb phasing of paretic and non-paretic limb during overground walking measured from biomechanical gait analysis.
Interlimb coordination in pedaling | Each training day, up to 24 times, through study completion which takes 6-8 weeks.
  Relative phasing of paretic and non-paretic limb during split-crank (i.e., bilateral uncoupled) pedaling calculated from position encoders coupled to right and left pedal.
Motorized intervention during pedaling split-crank (i.e., bilateral uncoupled) pedaling | Each training day, up to 24 times, through study completion which takes 6-8 weeks.
  Magnitude of assistance and resistance applied to the moving limbs during split-crank (i.e., bilateral uncoupled) pedaling measured as electrical current to the motors converted to units of torque.
Absences | Each day of training. There are 24 training sessions delivered over 6 weeks.
  Count the number times each participant misses a scheduled training session. Record the reason for the absence.
Adverse events | Each day of training. There are 24 training sessions delivered over 6 weeks.
  Count the number of adverse events, defined as any undesirable experience associated with CUped. Classify as mild, moderate, or severe. Classify by attribution as unrelated to protocol, possibly, probably, or definitely related to protocol.

SECONDARY OUTCOMES:
Muscle activity - timing | Pretest (1 day to 1 month before the intervention begins), Posttest (typically within 1 week of completing the intervention) and Midpoint of training (week 3)
  Recorded during pedaling with surface electrodes. Timing of EMG will be computed.
Muscle activity - amplitude | Pretest (1 day to 1 month before the intervention begins), Posttest (typically within 1 week of completing the intervention) and Midpoint of training (week 3)
  Recorded during pedaling with surface electrodes. Amplitude of EMG will be computed.
Physiological response to exercise - Blood pressure | Each training day, up to 24 times, through study completion which takes 6-8 weeks.
  Blood pressure (systolic and diastolic) in mm of Hg
Physiological response to exercise - Heart rate | Each training day, up to 24 times, through study completion which takes 6-8 weeks.
  Heart rate in beats per minute
Physiological response to exercise - Rate of perceived exertion | Each training day, up to 24 times, through study completion which takes 6-8 weeks.
  Rate of perceived exertion according to the Borg Scale. Scale range is 7-20 where larger values are more exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No